CLINICAL TRIAL: NCT03293537
Title: Skin Conductance and Heart Rate as Biomarkers to Uncover Covert Emotional Reactions in Patients With Dementia Associated Apathy; a Multi-centre Study.
Brief Title: Dementia Associated Apathy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Silke Neumann, MSc, Zurich University of Applied Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Biomarker and Apathy
Record Dates: First submitted 2017-09-21; First posted 2017-09-26 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Emotions; Dementia; Apathy
Keywords: Dementia; Aphathy; Emotion; Images; Skin conductance; Heart rate
MeSH Terms: conditions — Dementia; Lethargy | interventions — Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with dementia (Experimental): The subject will be informed of the procedure and their task before the sensors are attached. Electrodermal activity (EDA) and heart rate (HR) will be continuously monitored while the subject views the image sequence on a PC monitor. EDA will be measured using electrodes attached to the middle (D3) and ring finger (D4). Heart rate will be measured using an infrared pulseoximeter attached to one of the free digits of the hand. A pulseoximeter is a non-invasive sensor, using tissue absorption of infrared light to determine blood-oxygen saturation (SaO2). EDA and HR will be recorded concurrently using commercial software. Data analysis will involve both commercial and in-house software.
  Interventions: Diagnostic Test: Skin conductance and Heart rate measurement

INTERVENTIONS:
Diagnostic Test: Skin conductance and Heart rate measurement — while observing selected photos the Skin conductance and heart rate will be measured.

SUMMARY:
We want to determine if patients with dementia show any kind of emotion while they look at a defined selection of photos. These are photos taken from a international image-platform and mixed with photos (biographic) that show personal objects, personal events, etc.

While the photos will be presented each a few seconds the skin conductance and the heart rate will be measured. We want to find out if there is any emotion measurable while showing the photos.

DETAILED DESCRIPTION:
The lack of overt behaviour in individuals exhibiting dementia-associated apathy is not only stressful to family members and caregivers, it is also a major challenge for medical and nursing staff. Knowing whether apathy arises from an impaired function of the neural network of affect due to neurodegenerative processes accompanying dementia provides a neural explanation of this condition. Somatic indicators of affective responses (e.g., changes in skin conductance, or heart rate) are an effective means to uncover covert emotional responses in nursing home residents suffering from dementia associated apathy.

The overall objective is to determine whether dementia associated apathy is the result of an impaired functioning of the neural macro-network of affect. We want to compare the quantitative change in physiological parameters for each image category between individuals of the two subgroups: 1. Individual with dementia only and 2.individuals with dementia and dementia-associated apathy.

The primary objective is to uncover a covert emotional response using changes in skin conductance in patients with dementia and patients with dementia + dementia associated apathy.

The secondary objective is to uncover a covert emotional response using changes in the heart rate in patients with dementia and patients with dementia + dementia associated apathy.

Diagnosis of dementia, age at initial dementia diagnosis, age at initial apathy diagnosis, time since initial diagnosis of dementia and apathy will be obtained from medical records. The type and daily dose of medication as well as the type and frequency of occupational, physio- and psychosocial therapy will be drawn from medical records. The SMMSE (Severe Mini Mental State Examination)score will determine severity of dementia and the AES (Apathy Evaluation Scale )score the severity of apathy. Using the FAST (Functional Assessment Staging) will assess the capacity of performing the activities of daily life.

Measurements will be conducted in a familiar environment and in the presence of a family member or a member of staff to avoid any kind of stress and concern for the participant. The subject will be informed of the procedure and their task before the sensors are attached. Electrodermal activity (EDA) and heart rate (HR) will be continuously monitored while the subject views the image sequence on a PC monitor. EDA and HR will be recorded concurrently using commercial software. Data analysis will involve both commercial and in-house software. All data will be stored on a hard disk, in a compressed and encrypted format.

ELIGIBILITY:
Inclusion Criteria:

* existing medical diagnosis of dementia, independent of the presence or absence of neuropsychiatric symptoms.

We include nursing home residents with Informed Consent as documented by signature from the German speaking part of Switzerland with moderate to severe dementia.

The presence or absence of apathy serves to assign participants into the appropriate experiments group.

Exclusion Criteria:

* Known or suspected non-compliance, drug or alcohol abuse,

  * Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders
  * Previous enrolment into the current study,
  * Enrolment of the investigator, his/her family members, employees and other dependent persons,
  * Medically documented diagnosis of schizophrenia or bipolar disorder or the diagnosis of diminished intelligence.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Estimated)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Skin conductance | 15 minutes
  The change in skin conductance will be taken to be the peak amplitude of the change in skin conductance
Heart rate | 15minutes
  The heart rate measured in Hertz (HZ). The Heart rate will be measured using an infrared pulseoximeter attached to one of the free digits of the hand.

CONTACTS AND LOCATIONS:
Overall Officials: Heidrun Becker, Prof.DR., Study Chair — Zurich University of Applied Sciences
Locations (1):
- Zurich University of applied Sciences, Winterthur, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: No